CLINICAL TRIAL: NCT06351358
Title: A Multi-center, Open-label Study to Evaluate the Synergistic Effects of Biostimulator and Dermal Fillers for Cheek Augmentation and Correction of Contour Deficiencies
Brief Title: Evaluation of the Effects of a Biostimulator and Dermal Fillers for Cheek Augmentation and Contour Deficiencies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.036
Record Dates: First submitted 2024-03-20; First posted 2024-04-08 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Photoaging; Weight Loss; Skin Laxity; Photodamaged Skin; Volume Deficiency of the Midface
MeSH Terms: conditions — Weight Loss; Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Sculptra and Restylane Treatment Group (Experimental): Subjects in the treatment group will receive the intervention with Sculptra and Restylane Lyft or Restylane Contour.
  Interventions: Device: Sculptra treatment; Device: Restylane Treatment

INTERVENTIONS:
Device: Sculptra treatment — Subjects will receive treatment of Sculptra at baseline. Subjects will receive a second treatment of Sculptra at Week 4 visit. At the Week 8 visit, subjects will receive an optional treatment of Sculptra.
Device: Restylane Treatment — Subjects will receive treatment Restylane Lyft or Restylane Contour at baseline. Subjects will receive an optional touch-up of Restylane Lyft or Restylane Contour at Week 4 visit.

SUMMARY:
Adult subjects with a history of or currently taking glucagon-like peptide-1 (GLP-1) receptor agonist medication and moderate-to-severe cheek wrinkles and midface contour deficiencies will be treated with Sculptra correction of fine lines and wrinkles in the cheek area and Restylane Lyft or Restylane Contour for cheek augmentation and correction of midface contour deficiencies.

DETAILED DESCRIPTION:
This is a multi-center, open-label study. Subjects will be screened on the basis of the selection criteria for study qualification. Eligible subjects will have initial treatment of Sculptra and Restylane Lyft or Restylane Contour on both cheeks at the Baseline visit.

At Week 4, subjects will receive a second Sculptra treatment on both cheeks for optimal correction and an optional touch-up of Restylane Lyft or Restylane Contour for optimal correction, defined as at least a 1-grade improvement on the GCWS and MMVS.

At Week 8, subjects will receive an optional Sculptra treatment on both cheeks for optimal correction.

Subjects will have follow-up visits at Week 16, Week 28, and Week 40 if the last Sculptra treatment is at Week 4 or at Week 20, Week 32, and Week 44 if the last Sculptra treatment is at Week 8.

ELIGIBILITY:
Inclusion Criteria:

* Any Fitzpatrick skin types I-VI, with effort to include minimum n = 1 for each category per site
* Any races and ethnicities, with effort to include minimum n = 2 per site for whom identify as American Indian or Alaska Native, Eastern/Southeastern Asian, South Asians, Hispanic or Latino, Black or African American, Native Hawaiian or Other Pacific Islander, etc.
* Subject with moderate-to-severe cheek wrinkles on the GCWS
* Subject with mild-to-severe midface contour deficiencies on the MMVS
* Subject with intent to undergo correction of cheek augmentation or midface contour deficiencies.
* Subject with history of taking or currently taking GLP-1 receptor agonist medications such as semaglutide, liraglutide, etc.
* Subject with stable Body Mass Index (BMI) within 4-6 weeks before study start.
* Subject willing to maintain a stable Body Mass Index (BMI, ± 2 kg/m2) throughout the study.
* Willing to maintain the current lifestyle and daily routine (e.g., diet, exercise, sleep, etc.) throughout the study.
* Subject willing to be photographed at each visit.
* Subject willing to abstain from any other facial plastic surgical or cosmetic procedure(s) during the duration of the study.
* For female subjects of childbearing potential, she agrees to use an acceptable form of effective birth control for the duration of the study. Subjects must be willing to take a urine pregnancy test (UPT) prior to all treatments. (Females of non-childbearing potential, e.g., post-menopausal (absence of menstrual bleeding for 1 year without any other medical reason), hysterectomy, or bilateral ovariectomy, are not required to have a UPT.)
* Male subjects must be willing to shave prior to each study visit.
* Ability to read, understand and give consent for participation in the study.
* Agreement to adhere to the procedures and requirements of the study and to report to the site on the day(s) and at the time(s) scheduled for the assessments.

Exclusion Criteria:

* Pregnant, breastfeeding, or planning pregnancy during the course of the study.
* Current smokers or consumer of nicotine.
* History of allergy or hypersensitivity to any ingredient of the treatment products, anesthetics or lidocaine
* Previous or present multiple allergies or severe allergies, such as manifested by anaphylaxis or angioedema, or family history of these conditions
* Previous tissue-augmenting therapy, contouring, or revitalization treatment in the face, except the lips
* History of injectable polymethylmethacrylate (PMMA) treatment
* Previous treatment/procedure in the face in the previous 6 months that, in the Investigator's opinion, would interfere with the study injections and/or study assessments or exposed the study subject to undue risk by study participation, or planning to undergo any of these procedures in the treatment area at any time during the study
* Presence of any disease or lesions near or on the area to be treated
* History of bleeding disorders or treatment with anticoagulants or inhibitors of platelet aggregation (e.g., aspirin or other non-steroidal anti-inflammatory drugs), omega 3, or vitamin E within 14 days before treatment. Omega 3 and vitamin E are acceptable only as part of a standard multivitamin formulation.
* Previous surgery, including plastic surgery, lifting threads, tissue grafting, or tissue augmentation with permanent implants, silicone, tattoo affecting the treatment area, or any procedure, at the discretion of the Investigator, would interfere with the outcome of the study.
* Any medical condition that, in the opinion of the Investigator, would make the subject unsuitable for inclusion
* Other condition preventing the subject from entering the study in the Investigator's opinion
* Study site personnel, close relatives of the study site personnel (e.g., parents, children, siblings, or spouse), or employees and close relatives of employees at the Sponsor company.
* Participation in any interventional clinical study within 30 days of screening.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in skin hydration from baseline | Baseline, Week 4, Week 8, Week 16 or Week 20
  Corneometer (Courage + Khazaka, Germany) measurements will be taken in triplicate to assess skin hydration. The Corneometer measures in Corneometer units from 0 (no water at all) - 120 (on water).The locations of measurement will be at (1) the zygoma area in the Restylane-treated region using a ruler starting from the corner of the eye and (2) 2-3 cm laterally from the end of the earlobe in the Sculptra-injected region using a ruler starting from the end of the earlobe to the corner of the mouth. An increase in scores indicates an improvement.
Change in skin radiance from baseline | Baseline, Week 4, Week 8, Week 16 or Week 20
  Glossymeter (Courage + Khazaka, Germany) measurements will be taken to assess skin radiance. The results will be expressed in Glossymeter units. The locations of measurement will be at (1) the zygoma area in the Restylane-treated region using a ruler starting from the corner of the eye and (2) 2-3 cm laterally from the end of the earlobe in the Sculptra-injected region using a ruler starting from the end of the earlobe to the corner of the mouth. An increase in scores indicates an improvement.
Change in skin elasticity from baseline | Baseline, Week 4, Week 8, Week 16 or Week 20
  Cutometer (Courage + Khazaka, Germany) measurements will be taken to assess skin elasticity. The Cutometer measures skin elasticity in mm penetration depth per unit of time. The locations of measurement will be at (1) the zygoma area in the Restylane-treated region using a ruler starting from the corner of the eye and (2) 2-3 cm laterally from the end of the earlobe in the Sculptra-injected region using a ruler starting from the end of the earlobe to the corner of the mouth. An increase in scores indicates an improvement.
Change in skin thickness from baseline | Baseline, Week 4, Week 8, Week 16 or Week 20
  DermaLab® Ultrasound (Cortex Technology, Denmark) measurements will be taken in triplicate to assess skin thickness in µm. The locations of measurement will be at (1) the zygoma area in the Restylane-treated region using a ruler starting from the corner of the eye and (2) 2-3 cm laterally from the end of the earlobe in the Sculptra-injected region using a ruler starting from the end of the earlobe to the corner of the mouth. An increase in scores indicates an improvement.

SECONDARY OUTCOMES:
Subject Treatment Satisfaction | Week 4, Week 8, Week 16 or Week 20
  Subjects will be asked about their perception and satisfaction with the study treatments using a self-assessment questionnaire at each visit after Baseline. Questionnaires will be tabulated; and the frequency and percentage of all response options will be reported for each question and time point. Favorable responses (i.e., strongly agree and agree, yes), neutral responses (i.e., neither agree nor disagree, no difference), and unfavorable responses (i.e., strongly disagree and disagree, no) will be tabulated and reported as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Somenek, MD, Principal Investigator — Somenek + Pittman MD: Advanced Plastic Surgery; Paul Z Lorenc, MD, Principal Investigator — Z. Paul Lorenc Aesthetic Plastic Surgery
Locations (2):
- United States (2):
  - Somenek + Pittman MD: Advanced Plastic Surgery, Washington D.C., District of Columbia
  - Lorenc Aesthetic Plastic Surgery Center, New York, New York

IPD SHARING:
Plan to Share IPD: No